CLINICAL TRIAL: NCT05711277
Title: Comparison of the Taste and Acceptability of a New Ice Cream Based Supplement (Nottingham-Ice Cream) Compared to Standard Hospital Milkshake Oral Nutritional Supplement in Older Adults in Hospital Who Have Suffered a Broken Bone
Brief Title: The Taste and Acceptability of a High Protein Ice Cream Compared With Hospital Milkshake Nutritional Supplement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 22HC002
Record Dates: First submitted 2022-09-23; First posted 2023-02-02 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Femoral Fragility Fractures; Malnutrition
Keywords: Older adults; Malnutrition; Oral Nutritional Supplements; Fractures; Frailty; Dietary intake
MeSH Terms: conditions — Malnutrition; Fractures, Bone; Frailty | interventions — Dietary Supplements; Ice Cream

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N-ICE CREAM (Experimental)
  Interventions: Dietary Supplement: High protein, fortified, ice cream
- Milkshake ONS (Active Comparator)
  Interventions: Dietary Supplement: Standard milkshake ONS (Fortisip Compact Protein)

INTERVENTIONS:
Dietary Supplement: Standard milkshake ONS (Fortisip Compact Protein) — Two 125ml bottles of standard ONS administered a day for two days
  Other Names: ONS; Sip feeds; Oral nutritional supplements
  Arms: Milkshake ONS
Dietary Supplement: High protein, fortified, ice cream — Two 80g servings of N-ICE CREAM administered a day for two days
  Other Names: N-ICE CREAM; Nottingham-Ice cream
  Arms: N-ICE CREAM

SUMMARY:
This study aims to compare the acceptability of a new high protein, fortified, ice cream called Nottingham-Ice cream (N-ICE CREAM) with a standard milkshake-style oral nutritional supplement (ONS); Fortisip Compact Protein in older patients admitted to hospital with fractures who require ONS as part of routine care.

DETAILED DESCRIPTION:
Older adults admitted to hospital with fractures are often vulnerable to malnutrition. The European Society for Clinical Nutrition and Metabolism guidelines on clinical nutrition and hydration in geriatrics recommend 'older patients with hip fracture shall be offered ONS post-operatively to improve dietary intake and reduce risk of complications'.

As part of routine care at Nottingham University Hospitals (NUH) NHS Trust patients with femoral fragility fractures and vertebrae fractures are prescribed a milkshake style ONS called Fortisip Compact protein twice daily. Poor compliance (amount consumed relative to amount prescribed) to ONS in older adults has been reported in scientific literature with our own research findings reporting 28% compliance to standard milkshake ONS in older trauma and orthopaedic patients. There is a need for an ONS which patients accept and enjoy, of which ice cream has the strong possibility of accomplishing. There few studies to date exploring the potential of ice cream as a nutritional intervention. Ice cream has proven successful improving quality of life and shown favourable among oncological patients with 88% reporting they would rather eat ice cream that conventional nutritional supplements. Furthermore, research in ortho-geriatric patients at NUH showed an increase in energy intake by 41% for those consuming a high energy and protein ice cream. These encouraging results highlight the need for further scientific research to explore ice cream as an ONS.

This study aims to further explore compliance to N-ICE CREAM compared to standard ONS. This is a randomised crossover study. Participants admitted to hospital with hip or spine fractures and requiring ONS for the duration of their hospital stay only as part of routine care will receive N-ICE CREAM for two days and standard ONS for two days in a random order. Participants will complete acceptability and attitudes questionnaire for each product in additional to a questionnaire about the feasibility of having N-ICE CREAM at home. Compliance to each product will also be monitored and preference noted.

Overview of the study:

1. Patients will be assessed for inclusion and exclusion criteria by the research team, and then provided with information about the study. Patients eligible to take part will be asked for written informed consent or nominated consultee consent sought from patients without capacity. Participant demographics and medical history will be collected from online hospital systems and medical notes.
2. Participants will be randomly allocated to receive either:

A. N-ICE CREAM twice a day for two days; N-ICE CREAM tub size approximately 80g (1.96kcal/g, 0.19g protein/g) followed by a standard milkshake based ONS; Fortisip Compact Protein twice a day for two days; serving size 125ml (2.4kcal/g, 0.14g protein/g).

B. A standard milkshake based ONS; Fortisip Compact Protein twice a day for two days followed by N-ICE CREAM twice a day for two days.

The hypothesis is that N-ICE CREAM will be 'as accepted', if not more accepted, than the milkshake ONS. The results from this study will guide future nutritional interventions for older adults admitted to hospital with fractures.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years and over admitted to QMC hospital.
* Patients capable of giving informed consent, or if appropriate, participants having a personal consultee able to complete a declaration in favour of the patient participating in the trial.
* Patients with a diagnosed hip or spine fracture requiring ONS as part of the routine nutritional pathway.
* Patients who have had malnutrition risk assessed by the Malnutrition Universal Screening Tool (MUST) and have a MUST score of 0 or 1.
* Patients with an anticipated length of stay ≥ 4 days.

Exclusion Criteria:

* Patients < 65 years old.
* Patients scheduled for total parenteral nutrition or tube feeding.
* Patients with a MUST ≥ 2.
* Clinically unstable patients (e.g. in terminal condition end of life situation).
* Patients with medical or dietary contraindication to any feed ingredients (e.g. with known allergies or intolerance to any ingredients in the N-ICE CREAM or FSCP).
* Patients with significant renal impairment (chronic kidney disease stages 4 and 5).
* Any contraindication against nutritional therapy (includes paralytic ileus< inborn errors of metabolism of nutrients contained in N-ICE CREAM or FSCP).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of acceptability by questionnaire (taste, texture, aroma, consistency etc). | 4 days
  Questionnaire used to ask patients to rate sensory characteristics including appearance, taste/flavour, texture/consistency aroma/smell, taste/sweetness from dislike a lot to like a lot. The average of these scores will represent "overall acceptability." Questionnaire to be completed for Nottingham-Ice cream and the milkshake oral nutritional supplement.
  Dislike a lot = 1, dislike moderately = 2, dislike a little = 3, like a little = 5, like moderately = 6, like a lot = 7.
  Questionnaires will be undertaken on day two and four.
Evaluation of product preference | 4 days
  A single question questionnaire used to ask patients whether they preferred Nottingham-Ice cream or the milkshake oral nutritional supplement.

SECONDARY OUTCOMES:
Evaluation of compliance | 4 days
  Record daily the amount of Nottingham-Ice cream and milkshake oral nutritional supplement consumed by patients compared to the amount prescribed by either weighing waste, or from and estimated recall from patient or nursing staff.
  Good compliance = > 80% of being consumed.
Attitudes towards long term use of milkshake oral nutritional supplement and Nottingham-Ice cream by questionnaire | 4 days
  A questionnaire will be used to record confidence, from very unconfident to very confident, in being able to consuming each product over different time periods (two, four and twelve weeks) and maximum dose tolerated. The average score will represent "overall confidence."
  Very unconfident = 1, unconfident =2, confident = 4, very unconfident = 5.
  Questionnaires will be undertaken on day two and four.
Feasibility of having Nottingham-Ice cream at home | 4 days
  Patients to complete the 'Nottingham-Ice cream Feasibility at home' questionnaire. Questions will cover freezer accessibility and storage space, likelihood to store Nottingham-Ice cream and preferred ice cream tub size for storage.
  Questionnaire to be completed after patients have trialled Nottingham-Ice cream.

CONTACTS AND LOCATIONS:
Locations (1):
- Queens Medical Centre, Nottingham, Nottinghamshire, United Kingdom